CLINICAL TRIAL: NCT07298018
Title: A Pilot Study of RISE for Nurse Managers Retreat
Brief Title: RISE for Nurse Managers Retreat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2365808
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Burnout, Secondary Traumatic Stress, Perceived Stress
MeSH Terms: conditions — Burnout, Psychological; Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant group (Experimental): Intervention group will attend the RISE Retreat program, which is a 2.5-day retreat-style psychoeducational group program facilitated by licensed mental health professionals (LMHPs)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Psychoeducational group program designed to impact occupational and psychological indicators including resilience, insight, self-compassion, empowerment, burnout and secondary trauma

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of the RISE for Nurse Managers retreat and its impact on occupational and psychological well-being indicators

DETAILED DESCRIPTION:
The RISE program is an empirically supported wellbeing intervention for nurses and nurse leaders delivered over 8 or 9 weeks in 90-minute weekly sessions facilitated by a licensed mental health professional. The program themes are Resilience, Insight, Self-Compassion, and Empowerment. This study will be to examine the feasibility and acceptability of delivering the program in a retreat style format over 2.5 days.

ELIGIBILITY:
Inclusion Criteria:

* an employed AdventHealth Nurse Manager
* a "moderate" or "high" score in burnout equal to ≥17 in the Emotional Exhaustion Domain and/or ≥7 in the Depersonalization Domain on the MBI

Exclusion Criteria:

* a direct care RN, Nurse Director, Educator, and Executive
* a "low" score in burnout equal to <17 in the Emotional Exhaustion domain and/or <7 in the Depersonalization domain on the MBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Inventory - Human Services Survey | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  22-item questionnaire with the following response categories: 0=never, 1=a few times a year or less, 2=once a month or less, 3=a few times a month, 4=once a week, 5=a few times a week, 6=every day

SECONDARY OUTCOMES:
Professional Quality of Life Scale | Baseline, 1- and 3-and 6-month follow-up
  30-item questionnaire with the following response categories: 1=never, 2=rarely, 3=sometimes, 4=often, 5=very often
Brief Resilience Scale | Baseline, 1- and 3-and 6-month follow-up
  6-item questionnaire with the following response categories: 1=strongly agree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree
Self-Reflection and Insight Scale | Baseline, 1- and 3-and 6-month follow-up
  20-item questionnaire with the following response categories: 1=strongly disagree, 2, 3, 4, 5, 6=strongly agree
Self-Compassion Scale Short Form | Baseline, 1- and 3-and 6-month follow-up
  12-item questionnaire with the following response categories: 1=almost never, 2, 3, 4, 5=almost always
General Self-Efficacy Scale | Baseline, 1- and 3-and 6-month follow-up
  10-item questionnaire with the following response categories: 1=not at all true, 2=barely true, 3=moderately true, 4=exactly true
Perceived Stress Scale | Baseline, 1- and 3-and 6-month follow-up
  10-item questionnaire with the following response categories: 0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often
Generalized Anxiety Disorder - 2 item scale | Baseline, 1- and 3-and 6-month follow-up
  2-item questionnaire with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day
Patient Health Questionnaire - 2 item | Baseline, 1- and 3-and 6-month follow-up
  2-item scale with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day
Post-Traumatic Growth Inventory | Baseline, 1- and 3-and 6-month follow-up
  21-item scale scored using six-point responses: zero ("I did not experience this change as a result of my crisis") to five ("I experienced this change to a very great degree as a result of my crisis")
Psychological Empowerment Instrument | Baseline, 1- and 3-and 6-month follow-up
  12-item measure that assesses empowerment in the workplace using a 7-point Likert response scale. Four aspects are measured: meaning, competence, self-determination, and impact.
Employment Status | 12-month post-program
  Human Resources Data

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T. Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey AK, Sawyer AT, Robinson PS. A Psychoeducational Group Intervention for Nurses: Rationale, Theoretical Framework, and Development. J Am Psychiatr Nurses Assoc. 2023 May-Jun;29(3):232-240. doi: 10.1177/10783903211001116. Epub 2021 Jun 22. PMID 34154451
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Litz BT, Plouffe RA, Nazarov A, Murphy D, Phelps A, Coady A, Houle SA, Dell L, Frankfurt S, Zerach G, Levi-Belz Y; Moral Injury Outcome Scale Consortium. Defining and Assessing the Syndrome of Moral Injury: Initial Findings of the Moral Injury Outcome Scale Consortium. Front Psychiatry. 2022 Jul 5;13:923928. doi: 10.3389/fpsyt.2022.923928. eCollection 2022. PMID 35873252
- [Background] Maslach C, Jackson SE, Leiter MP. Maslach Burnout Inventory manual, 3rd ed. Palo Alto, CA: Consulting Psychologists Press, 1996.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Sawyer AT, Bailey AK, Green JF, Sun J, Robinson PS. Resilience, Insight, Self-Compassion, and Empowerment (RISE): A Randomized Controlled Trial of a Psychoeducational Group Program for Nurses. J Am Psychiatr Nurses Assoc. 2023 Jul-Aug;29(4):314-327. doi: 10.1177/10783903211033338. Epub 2021 Jul 23. PMID 34293934
- [Background] Sawyer AT, Tao H, Bailey AK. The Impact of a Psychoeducational Group Program on the Mental Well-Being of Unit-Based Nurse Leaders: A Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Jun 2;20(11):6035. doi: 10.3390/ijerph20116035. PMID 37297639
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy Scale. J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs, 35, 37.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spreitzer GM. Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal. 1995; 38(5):1442-1465.
- [Background] Stamm, B. H. (2010). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL). http://www.proqol.org.
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649